CLINICAL TRIAL: NCT03279458
Title: Non-invasive Tidal Volume Monitoring Using the Linshom Respiratory Monitoring Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Madhankumar Sathyamoorthy, Associate Professor, University of Mississippi Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-0063
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Results first posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Pulmonary Ventilation; Capnography
Keywords: Capnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Linshom Respiratory Monitoring Device (Experimental): Volunteers will breathe through a continuous positive airway pressure (CPAP) face mask fitted with the Linshom device. The volunteers will be instructed to breathe normal through the CPAP mask on room air. The excursions of the thermistor tracings (from valley to peak) will be recorded by the Linshom device and displayed continuously on a laptop monitor in a waveform.
  Interventions: Device: Linshom Respiratory Monitoring Device
- Ventilator (Active Comparator): Volunteers will breathe through a continuous positive airway pressure (CPAP) face mask fitted with the Linshom device. The volunteers will be instructed to breathe normal through the CPAP mask on room air.The tidal volume will also be measured by the ventilator and the data downloaded in a Compact Flash card.
  Interventions: Device: Linshom Respiratory Monitoring Device

INTERVENTIONS:
Device: Linshom Respiratory Monitoring Device — Volunteers will breathe through a continuous positive airway pressure (CPAP) face mask fitted wth the Linshom device. The volunteers will be instructed to breathe normal through the CPAP mask on room air. The excursions of the thermistor tracings (from valley to peak) will be recorded by the Linshom device and displayed continuously on a laptop monitor in a waveform. The tidal volume will also be measured by the ventilator and the data downloaded in a Compact Flash card.

SUMMARY:
Many post-operative complications arise from patients who breathe inadequately. Inadequate respiration, whether the result of surgery or the anesthesia, causes a decrease in blood oxygen saturation and an increase in carbon dioxide partial pressure. Both of these surrogate measurements of respiration may pose a challenge to measure. Some administer exogenous oxygen to all patients as they leave the operating room in order to maintain the blood oxygen saturation. This renders the oximeter a less sensitive metric of depressed respiration. In the face of decreased respiration, the carbon dioxide levels continue to increase slowly and often go undetected unless blood gases are measured. Indeed carbon dioxide blood levels are the only metric to detect inadequate ventilation using this surrogate index.

Monitoring ventilation is a serious challenge outside of critical care settings. In fact, there are no monitors available that can measure tidal volume or relative tidal volume outside of these settings.

Linshom is a novel instrument that tracks relative respiration by measuring the excursions of the temperature swings between inspiration and expiration and normalizing them to the patient's breathing. This monitor may be the first non-invasive monitor to measure relative tidal volume in non-critical care settings.

The purpose of this study is to determine whether a non-invasive, temperature-based respiratory instrument can track tidal volume (Vt) in patients.

The investigators hypothesize that the Linshom device can accurately and consistently track tidal volume as measured by closed loop mechanical ventilator.

DETAILED DESCRIPTION:
Forty volunteers will be enrolled in this open label, prospective study to determine the correlation between the tidal volumes measured with the Linshom detector and those measured with the mechanical ventilator. after Institutional Review Board (IRB) approval and written informed consent from the volunteers.

The Linshom detector, which is comprised of two rapid responding medical-grade thermistors in close proximity to the mouth/nose (sensor) and a thermistor remote to the airway, will be mounted in the continuous positive airway pressure (CPAP) face mask to measure the temperature during breathing. The CPAP will be connected to a Servo-I ventilator (Maquet) with a circuit and disposable filter. The volunteers will be instructed to breathe normal through the CPAP mask on room air. The excursions of the thermistor tracings (from valley to peak) will be recorded by the Linshom device and displayed continuously on a laptop monitor in a waveform. The tidal volume will also be measured by the ventilator and the data downloaded in a Compact Flash card. The temperature profiles from the sensors and the relative tidal volume will be correlated with the tidal volumes measured by the ventilator.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* pregnant
* suffer from claustrophobia
* had recent respiratory illness
* had recent gastrointestinal illness
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhankumar Sathyamoorthy, MBBS, MS, Principal Investigator — Children's of Mississippi/University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Background] Manifold CA, Davids N, Villers LC, Wampler DA. Capnography for the nonintubated patient in the emergency setting. J Emerg Med. 2013 Oct;45(4):626-32. doi: 10.1016/j.jemermed.2013.05.012. Epub 2013 Jul 18. PMID 23871325
- [Background] Brouillette RT, Morrow AS, Weese-Mayer DE, Hunt CE. Comparison of respiratory inductive plethysmography and thoracic impedance for apnea monitoring. J Pediatr. 1987 Sep;111(3):377-83. doi: 10.1016/s0022-3476(87)80457-2. PMID 3625404
- [Background] Ramsay MA, Usman M, Lagow E, Mendoza M, Untalan E, De Vol E. The accuracy, precision and reliability of measuring ventilatory rate and detecting ventilatory pause by rainbow acoustic monitoring and capnometry. Anesth Analg. 2013 Jul;117(1):69-75. doi: 10.1213/ANE.0b013e318290c798. Epub 2013 Apr 30. PMID 23632055
- [Background] Keidan I, Gravenstein D, Berkenstadt H, Ziv A, Shavit I, Sidi A. Supplemental oxygen compromises the use of pulse oximetry for detection of apnea and hypoventilation during sedation in simulated pediatric patients. Pediatrics. 2008 Aug;122(2):293-8. doi: 10.1542/peds.2007-2385. PMID 18676546
- [Background] Williamson JA, Webb RK, Cockings J, Morgan C. The Australian Incident Monitoring Study. The capnograph: applications and limitations--an analysis of 2000 incident reports. Anaesth Intensive Care. 1993 Oct;21(5):551-7. doi: 10.1177/0310057X9302100510. PMID 8273874
- [Background] Nassi N, Piumelli R, Lombardi E, Landini L, Donzelli G, de Martino M. Comparison between pulse oximetry and transthoracic impedance alarm traces during home monitoring. Arch Dis Child. 2008 Feb;93(2):126-32. doi: 10.1136/adc.2007.118513. Epub 2007 Sep 24. PMID 17893118
- [Background] Kasuya Y, Akca O, Sessler DI, Ozaki M, Komatsu R. Accuracy of postoperative end-tidal Pco2 measurements with mainstream and sidestream capnography in non-obese patients and in obese patients with and without obstructive sleep apnea. Anesthesiology. 2009 Sep;111(3):609-15. doi: 10.1097/ALN.0b013e3181b060b6. PMID 19672177
- [Background] Lerman J, Feldman D, Feldman R, Moser J, Feldman L, Sathyamoorthy M, Deitch K, Feldman U. Linshom respiratory monitoring device: a novel temperature-based respiratory monitor. Can J Anaesth. 2016 Oct;63(10):1154-1160. doi: 10.1007/s12630-016-0694-y. Epub 2016 Jul 13. PMID 27412466
- See also: A thermodynamic breathing sensor - a new non-invasive monitor of respiration — http://www.asaabstracts.com/strands/asaabstracts/abstract.htm%20%20;jsessionid=682567A35143EC5A44D16DFEEE86493A?year=2015&index=8&absnum=4494

RESULTS

PARTICIPANT FLOW:
Groups:
- Linshom Respiratory Monitoring Device: Volunteers will breathe through a continuous positive airway pressure (CPAP) face mask fitted with the Linshom device. The volunteers will be instructed to breathe normal through the CPAP mask on room air. The excursions of the thermistor tracings (from valley to peak) will be recorded by the Linshom device and displayed continuously on a laptop monitor in a waveform. The tidal volume will also be measured by the ventilator and the data downloaded in a Compact Flash card.
Period: Overall Study
Arm/Group | Linshom Respiratory Monitoring Device
Started | 40
Completed (The milestone was met if the participant was able to complete the breathing exercise.) | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Linshom: Linshom Respiratory Monitoring Device: Volunteers will breathe through a continuous positive airway pressure (CPAP) face mask fitted wth the Linshom device. The volunteers will be instructed to breathe normal through the CPAP mask on room air. The excursions of the thermistor tracings (from valley to peak) will be recorded by the Linshom device and displayed continuously on a laptop monitor in a waveform. The tidal volume will also be measured by the ventilator and the data downloaded in a Compact Flash card.
Arm/Group | Linshom
Number analyzed (Participants) | 40
Age, Customized [Count of Participants; unit: Participants]
  >= 18 years | 40
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The sex of participants was not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40
Number of participants [Count of Participants; unit: Participants] | 40

OUTCOME MEASURES:

1. Primary Outcome: Tidal Volume of Each Breath Was Measured Using the Same Breathing Mask CPAP Apparatus Combined With Respiratory Monitoring Device Allowing for Simultaneous Recording.
Description: Tidal volume measured by CPAP mask with Lishom respiratory monitoring device. Tidal volume determined from the ventilator will be compared to tidal volume measured by Linshom (calculated indirectly by temperature changes by computer algorithm)
Time Frame: 5 minutes
Population: Thirty participants successfully completed the experiment, which involved breathing through a CPAP mask in order to have the Linshom device record excursions of the thermistor tracings while the ventilator concurrently measured tidal volume.
Measure: Least Squares Mean (95% Confidence Interval); unit: ml
Groups:
- Maquet Ventilator: Tidal volume measured by the Maquet ventilator connected to CPAP mask concurrently with Linshom
Arm/Group | Linshom | Maquet Ventilator
Number analyzed (Participants) | 30 | 30
ml | 0.94 [0.88 to 0.97] | 0.94 [0.88 to 0.97]
Statistical Analysis 1: Comparison: Linshom vs Maquet Ventilator; Test type: Other — least square regression analysis; p < 0.05, Regression, Linear; correlation coefficient (R) = 0.94, 95% CI 2-sided [0.88 to 0.97]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for approximately 30 minutes, including the time while the patient was using the mask and the time immediately after completing the study.
Groups:
- Linshom: Linshom Respiratory Monitoring Device: Volunteers will breathe through a continuous positive airway pressure (CPAP) face mask fitted wth the Linshom device. The volunteers will be instructed to breathe normal through the CPAP mask on room air. The excursions of the thermistor tracings (from valley to peak) will be recorded by the Linshom device and displayed continuously on a laptop monitor in a waveform.
- Maquet Ventilator: The tidal volume will also be measured by the maquet ventilatorconcurrently and the data downloaded in a Compact Flash card.
Arm/Group | Linshom | Maquet Ventilator
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT03279458/Prot_SAP_001.pdf